CLINICAL TRIAL: NCT02709031
Title: Cicletanine in Hypertension With Diabetes: Added Magnesium Preserves Potassium and Sodium
Acronym: CHAMP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Navitas Pharma (Industry)
Collaborators: IndiPharm Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAV-011
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Arterial Hypertension; Diabetes; Hypokalemia; Hyponatremia
Keywords: Cicletanine; Magnesium; Metabolic disease
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Hypokalemia; Hyponatremia; Metabolic Diseases | interventions — cicletanine; Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cicletanine (Active Comparator): Patients will take escalating doses of cicletanine
  Interventions: Drug: Cicletanine
- Cicletanine + magnesium (Experimental): Patients will take escalating doses of cicletanine; patients will in addition take magnesium
  Interventions: Drug: Cicletanine + magnesium

INTERVENTIONS:
Drug: Cicletanine + magnesium — Cicletanine is an orally-dosed furopyridine drug launched or hypertension in France in 1988 (and soon thereafter in Germany by IPSEN. While the drug's maximum tolerated dose is not known, the principal concern (and so far only material concern) at higher doses is the decrease in levels of sodium and potassium. Trials so far have take n the drug up to 400 mg QD (once daily); it was well tolerated at that dose. The drug has had an excellent safety profile in its ~1.8 million patient-years of post-launch experience,
  Magnesium is being added to cicletanine in order to decrease losses of potassium and sodium, thereby enhancing cicletanine's safety at higher doses.
  Arms: Cicletanine + magnesium
Drug: Cicletanine — Cicletanine is an orally-dosed furopyridine drug launched or hypertension in France in 1988 (and soon thereafter in Germany by IPSEN. While the drug's maximum tolerated dose is not known, the principal concern (and so far only material concern) at higher doses is the decrease in levels of sodium and potassium. Trials so far have take n the drug up to 400 mg QD; it was well tolerated at that dose. The drug has had an excellent safety profile in its ~1.8 million patient-years of post-launch experience,
  Arms: Cicletanine

SUMMARY:
Cicletanine, which has been approved and launched for hypertension in France and Germany, has promise beyond hypertension in critically-unmet needs such as diabetes. It is evident from in vitro, animal and human studies that cicletanine's optimal dose in diabetes and other challenging, critically-unmet needs is likely to be higher than that for hypertension. Cicletanine's maximum tolerated dosage is not known, but the drug's dose-limiting effects are documented to be potassium loss and sodium loss from thiazide-type activity (one of the therapeutic mechanisms the drug is known to have); such thiazide-type losses are known to be reversed safely by magnesium. This trial explores the ability of magnesium to enhance cicletanine safety at higher doses in a trial involving patients with hypertension complicated by diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Sitting SBP (systolic blood pressure) > 150 mmHg (millimeters of mercury) after five minutes' rest.
2. Type II diabetes, with HbA1c between 8.5 and 11.5%. If a patient at screening presents outside of this range, the investigator may elect to re-screen a patient once to determine further the patient's eligibility.
3. Age >18 and < 80 years of age
4. BMI between 20 and 35, inclusive
5. Have been stable on existing therapy for at least 30 days prior to initiation of cicletanine (Visit 2)

   a. no change in antihypertensive nor antihyperglycemia agent dose within 30 days prior to screening visit.
6. Willing to comply with the requirements of the protocol.
7. Willing to provide written Informed Consent to participate in the study approved by an appropriately constituted IRB (Institutional Review Board).
8. All females who are not post-menopausal should be using at least two forms of contraception during the entire study.

Exclusion Criteria:

1. Use of potassium supplementation over the past 30 days
2. Use of potassium-wasting diuretics, e. g., thiazides over the past 30 days
3. AST (aspartate aminotransferase; also abbreviated SGOT) outside normal range of 5 and 40 mg/dL inclusive
4. ALT (alanine aminotransferase; also abbreviated SGPT) outside normal range of 7 and 56 mg/dL inclusive
5. Laboratory findings outside of normal range can be considered grounds for exclusion at the discretion of the Sponsor, Medical Monitor and / or Principal Investigator
6. History of or positive laboratory test for HIV, HBV (hepatitis B virus) or HCV (hepatitis C virus)
7. Clinically significant psychiatric, addictive or neurologic disease or any other condition that, in the Investigator's opinion, would compromise his/her ability to give informed consent, participate fully in this study, or prevent adherence to the requirements of the study protocol
8. Evidence of unstable cardiovascular disease including intermittent atrial fibrillation or unstable angina within the 4 weeks prior to screening
9. History of myocardial infarction, coronary artery bypass graft surgery, or percutaneous cardiac intervention within the last 3 months
10. Clinically significant valvular heart disease in the opinion of the Investigator
11. History of cerebrovascular accident or transient ischemic attack within the last 3 months
12. Presence or history of malignancy that required significant medical intervention within the preceding 3 months and/or is likely to result in death within the next 2 years
13. Chronic renal impairment or renal insufficiency defined by a serum creatinine ³ 2.5 mEq/dL and/or the requirement for dialysis
14. The subject is lactating, breastfeeding, or pregnant
15. The subject has received any investigational medication within 30 days prior to the start of this study or be scheduled to receive another investigational drug during the course of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Time to potassium rescue | 13 weeks (duration of study)
  The primary endpoint is the preservation of potassium levels at or above 3.3 mEq/L (milliequivalents per liter). A time to event model using the Log Rank test will be used to compare the Mg Group and those in the Non-Mg Group.

SECONDARY OUTCOMES:
Reduction in systolic blood pressure vs. baseline | 13 weeks (duration of study)
  Aggregate measure made for all 24 patients (12 cicletanine + magnesium; 12 cicletanine only). Subgroup analyses will also be made as feasible.
Reduction in diastolic blood pressure vs. baseline | 13 weeks (duration of study)
  Aggregate measure made for all 24 patients (12 cicletanine + magnesium; 12 cicletanine only). Subgroup analyses will also be made as feasible.
Reduction in HbA1c vs. baseline | 13 weeks (duration of study)
  Aggregate measure made for all 24 patients (12 cicletanine + magnesium; 12 cicletanine only). Subgroup analyses will also be made as feasible.
CRP (C reactive protein) levels | 13 weeks (duration of study)
  CRP (C-reactive protein) is a measure of general inflammation.
  This will be an aggregate measure made for all 24 patients (12 cicletanine + magnesium; 12 cicletanine only). Subgroup analyses will also be made as feasible.
Average levels of potassium in patients on cicletanine with and without magnesium | 13 weeks (duration of study)
  The average potassium levels levels in the two groups (cicletanine + magnesium; cicletanine only) will be compared. Subgroup analyses will also be made as feasible.
Average levels of sodium in patients on cicletanine with and without magnesium | 13 weeks (duration of study)
  The average sodium levels levels in the two groups (cicletanine + magnesium; cicletanine only) will be compared. Subgroup analyses will also be made as feasible.
Average levels of magnesium in patients on cicletanine with and without magnesium | 13 weeks (duration of study)
  The average magnesium levels levels in the two groups (cicletanine + magnesium; cicletanine only) will be compared. Subgroup analyses will also be made as feasible.

IPD SHARING:
Plan to Share IPD: No